CLINICAL TRIAL: NCT02911402
Title: Evaluation and Characterization of Motion Sickness on Passengers Sailing on the Astrolabe
Brief Title: Motion Sickness on Astrolabe's Vessel
Acronym: SICKVEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 14-153
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Sea Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: sea sickness questionnaires

SUMMARY:
Sea sickness syndrome is present for 80% of persons on board when the boat rotation missions Astrolabe, sometimes there is a risk of very significant dehydration. A special unit specialized in the fundamental study of the vestibular system (inner ear), sensory organ at the base of visual-vestibular conflict inducing this syndrome, also provides medical support for parabolic flights (flight reproducing weightlessness) where this syndrome is strongly present. The goal of the study is to assess the frequency of occurrence of this sea sickness syndrome on the Astrolabe, to understand the triggers (type of boat movements, personality traits, anxiety / stress) without changing habits on board for those on board taking a antinaupathique treatment given by the ship's doctor. This study will be done in collaboration between INSERM U 1075 (France) and the Laboratory of military research VIPER specialized in extreme environments (Belgium). The ultimate goal will be to provide the best recommendations and the best treatment regimen to alleviate as best as possible the symptoms of people on board of the Astrolabe so scientists on board can perform their work.

DETAILED DESCRIPTION:
Background: The objectives were to assess the prevalence, severity, medication taken and to look for predictive factors, in order to better identify characteristics of passengers at risk of motion sickness during transport scientists travelling from Hobart in Tasmania to the French polar stations in Antarctica.

Methods: Two hundred and thirty-nine passengers were surveyed over 4 years with 4 round trips per year using Motion Sickness Susceptibility Questionnaire (MSSQ), Simulator Sickness Questionnaire (SSQ), state-trait anxiety test (STAI-Trait and STAI-State), and general parameters (age, gender, number of trips, jet-lag, direction of the trip), medication, calculation of the distance of each passenger's cabin to the Centre of Gravity (CoG.).

ELIGIBILITY:
Inclusion Criteria:

* participant aged of 18 or older but younger than 70 who received their medical ability to travel to Terre Adélie or making a research cruise aboard the Astrolabe
* particpant signing the informed consent.

Exclusion Criteria:

* none

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Astrolabe passengers
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2014-10; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Motion Sickness susceptibilty questionnaire (fMSSQ) | day 1 to day 10
  Sensitivity of motion sickness
STAY-YA questionnaire | day 1 to day 10
  anxiety
STAY-YB questionnaire | day 1 to day 10
  anxiety
Vis-Morgen Questonnaire about sleeping | day 1 to day 10
  Subjective sleep scoring
Fatigue questionnaire | day 1 to day 10
  Tiredness
Dietary intake survey | day 1 to day 10
  food intake

SECONDARY OUTCOMES:
type of movement from the ship using use the data from the Dynamic Positioning System on board | baseline and every day up to 10 days
  boat motion
data from individual actigraphs worn by the participants | baseline and every day up to 10 days
  this will allow to quantify particpant's movements related to the ship movement
personnality questionnaire (OCEAN) | baseline and every day up to 10 days
  Personnality
anxiety questionnaire (STAY). | baseline and every day up to 10 days
  anxiety
treatment taken (international denomination and dose) | baseline and every day up to 6 days
  treatment taken by subject for motion sickness

CONTACTS AND LOCATIONS:
Overall Officials: stephane Besnard, MD, Principal Investigator — CaenHU
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No